CLINICAL TRIAL: NCT00132938
Title: An Open-label, Randomized, Multicenter, Clinical Study to Compare the Effects of Telithromycin, Azithromycin and Cefuroxime Axetil on the Penicillin or Macrolide Resistance of Streptococcus Pneumoniae in Patients With Acute Exacerbation of Chronic Bronchitis
Brief Title: PERSPECTIVE: Telithromycin - Acute Exacerbation of Chronic Bronchitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A_4020; EudraCT # :2004-001412-30
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic | interventions — telithromycin

INTERVENTIONS:
Drug: telithromycin

SUMMARY:
Primary Objective:

* The primary objective of the study is to demonstrate the superiority of telithromycin over azithromycin and over cefuroxime axetil in the reduction of Streptococcus pneumoniae (Sp) strains resistant to beta-lactams or macrolides at the Test of Cure (TOC) visit in the sputum of patients with Sp detected at the start of the study (Visit 1).

Secondary Objectives:

The secondary objectives of the study are:

* To demonstrate the superiority of telithromycin over azithromycin and over cefuroxime axetil in achieving clinical cure and Sp eradication success at the Test of Cure visit in patients with Sp detected in sputum specimen at the start of the study (Visit 1);
* To compare the clinical cure rates achieved by each treatment group in the penicillin or erythromycin resistant Sp (PERSp) population with the cure rates in the sensitive Sp (SSp) population at the End of Therapy (EOT) and Test of Cure visits;
* To compare the effect of telithromycin, azithromycin and cefuroxime axetil at the End of Therapy visit on the presence of Streptococcus pneumoniae strains resistant to beta-lactams or macrolides in the sputum of patients with Sp detected at the start of the study (Visit 1);
* To compare the clinical efficacy at the End of Therapy visit and safety at the Test of Cure visit of telithromycin, azithromycin and cefuroxime axetil in the "global" randomized population.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following criteria will be considered for enrollment into the study:

* Outpatients, male or female, aged 35 years or older
* Patients with a documented history of chronic bronchitis, characterized by cough and excessive sputum production for most days of at least three months for 2 consecutive years
* Patients with a clinical diagnosis of acute exacerbation of chronic bronchitis (AECB), presumed due to bacterial infection based on increased sputum purulence with either increased dyspnea or sputum volume
* Patients producing spontaneous sputum
* Patients with three or less AECB in the previous 12 months

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study:

* Patients with a known diagnosis of bronchiectasis; cystic fibrosis; lung cancer or lung metastases; active pulmonary tuberculosis; or with suspected pneumonia.
* Patients with present acute respiratory failure or patients requiring aggressive airway management
* Hospitalized patients and patients from institutional care facilities
* Patients treated with antibiotics within 14 days prior to enrollment
* Patients who are receiving other medications, including systemic antimicrobial agents; or who have other disease conditions or infections that could interfere with the evaluation of drug efficacy or safety.
* Patients with a concomitant condition (including clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease) making either implementation of the protocol or interpretation of the study results difficult
* Patients with a progressively fatal disease, or life expectancy ≤ three months
* Patients who have received any other investigational drug within 1 month prior to study entry, or have such treatment planned for the study period
* Patients with a recent (within the previous three months) history of alcohol or drug abuse
* Immunocompromised patients including, but not limited to: patients with known HIV infection (CD4 + <200/mm3); known neutropenia (<1500 neutrophils/mm3); chronic corticosteroid therapy (≥ 10mg/day prednisolone equivalent during at least three months); immunodepressant treatment within the previous six months; splenectomized patients or patients with known hyposplenia or asplenia.
* Patients with mental conditions rendering them unable to understand the nature, scope, and possible consequences of the study
* Patients unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and are unlikely to complete the study
* Patients having received anti-pneumococcal immunization in the previous six months before study entry
* Patients with suspected or known hypersensitivity to, or suspected serious adverse reactions to the study medication, or to ß-lactams or macrolide classes of antibiotics
* Patients diagnosed with myasthenia gravis
* Women who are breast-feeding or who are pregnant
* Women who are of childbearing potential who do not agree to use an approved contraceptive method during the study
* Patients with galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Patients with a known history of long QTc syndrome (e.g., personal or family history of syncope or arrhythmia)
* Patients treated within 2 weeks prior to study entry, or requiring treatment during study medication, with CYP3A4 inducers such as rifampicin, phenytoin, carbamazepine, phenobarbital, and St John's wort
* Patients requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Patients known to have impaired hepatic function
* Patients known to have impaired renal function
* Patients already enrolled in this study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5660
Dates: Start 2004-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Presence of PERSp in sputum of patients at the TOC visit in each treatment group and who were Sp positive in sputum at Visit 1.

SECONDARY OUTCOMES:
Assessment of clinical signs and symptoms of AECB at EOT visit for the global efficacy analysis population & at TOC visit for patients who were Sp positive in sputum at visit 1.Bacteriological data at EOT and TOC visits. Assessment of safety...

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Perdriset, MD, Study Director — Sanofi
Locations (8):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Budapest, Hungary
- Sanofi-Aventis, Casablanca, Morocco
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Mégrine, Tunisia
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)